CLINICAL TRIAL: NCT06139315
Title: A Single-blind, Randomised, Placebo-controlled, Parallel Group Design Phase I Trial to Investigate the Safety, Tolerability and Pharmacokinetics of Different Doses (Part A) and Different Treatment Regimens (Part B) of BI 765845 Administered to Healthy Male Subjects and Female Subjects of Non-childbearing Potential
Brief Title: A Study to Test How Well Different Doses of BI 765845 Are Tolerated by Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1478-0001; 2021-004733-36 (EudraCT Number)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BI 765845 treatment group (Part A) (Experimental): Part A
  Interventions: Drug: BI 765845
- BI 765845 treatment group (Part B) (Experimental): Part B
  Interventions: Drug: BI 765845
- Placebo group (Placebo Comparator): Part A and B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 765845 — BI 765845
  Arms: BI 765845 treatment group (Part A); BI 765845 treatment group (Part B)
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 765845 in healthy male subjects and female subjects of non-childbearing potential following intravenous administration of single rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive). Subjects should have a minimum bodyweight of at least 50 kg (inclusive).
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Male subject, who meets any of the following criteria for a highly effective contraception from at least screening until at least 90 days after drug administration:

  * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal) by female woman of childbearing potential (WOCBP) partner, plus condom in male subject
  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants) by female WOCBP partner, plus condom in male subject
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS) by female WOCBP partner, plus condom in male subject
  * Male subject is sexually abstinent
  * Male subject is vasectomised (vasectomy at least 1 year prior to enrolment) and received medical assessment of the surgical success (documented absence of sperm)
  * Female partner is surgically sterilised (including hysterectomy)
  * Female partner is postmenopausal, defined as no menses for at least 1 year without an alternative medical cause (in questionable cases a blood sample with follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory, if available) or
  * Female subject of non-childbearing potential, who meets any of the following criteria:

    * Female subject is surgically sterilised (including hysterectomy)
    * Female subject is postmenopausal, defined as no menses for at least 1 year without an alternative medical cause (in questionable cases a blood sample with FSH above 40 U/L and estradiol below 30 ng/L at screening is confirmatory)
* Male subjects are required to use condoms to prevent unintended exposure of their partner (both, male and female) to the trial drug via seminal fluid and should therefore use a condom at least from time point of administration of trial medication until completion of the trial. Alternatively, true abstinence is acceptable, if it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active, but becomes active with their partner, they must comply with the contraceptive requirements detailed above. Male subjects should not donate sperm for the duration of the trial until at least 90 days after drug administration.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders (including any history of cardiovascular diseases such as atherosclerosis, previous myocardial infarction or angina pectoris)
* Diseases of the central nervous system (including but not limited to any kind of seizures or history of stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant chronic or acute infections
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events | Up to 73 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in serum over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to Day 71
Maximum measured concentration of the analyte in serum (Cmax) | Up to Day 71

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com